CLINICAL TRIAL: NCT03200457
Title: Comparison of the Variability of Hepatic Load Quantification in Iron and Fat Estimated by MRI at 1.5 and 3 Tesla
Acronym: HEMOCOMPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-A01291-52
Record Dates: First submitted 2017-06-22; First posted 2017-06-27 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Iron Hepatic Overload; Fat Hepatic Overload
Keywords: Liver iron; Liver steatosis; MRI
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with hepatic iron overload or steatosis (Experimental): Each patient (80) will have two MRI exams on the same day: one performed in common practice on a 1.5 Tesla device and the other on a 3 Tesla device.
  Interventions: Device: 1,5 Tesla abdominal MRI; Device: 3 Tesla abdominal MRI

INTERVENTIONS:
Device: 1,5 Tesla abdominal MRI — Measurement of the fat and iron
Device: 3 Tesla abdominal MRI — Measurement of the fat and iron

SUMMARY:
The study proposes to compare the results of two examinations at 1.5 and 3 Tesla obtained on the same day on a series of 80 patients.

DETAILED DESCRIPTION:
Quantification of hepatic iron by MRI is validated at 1.5 Tesla on a small number of subjects with some discrepancies between the two most used techniques (liver to muscle ratio or calculation of the decay rate of the T2 * signal). Since the initial publications at 1.5 Tesla, new technical innovations have emerged which can allow better quantification. Recently, the investigators have applied these innovations to Rennes and have validated (SURFER study) the possibility of making a quantification of iron and fat on two 3 Tesla devices with good results in a single apnea acquisition. But it is not uncommon to have, in a structure, different magnetic field devices, and it is important to ensure that the results are transposable. It is also crucial for multicentre or cohort studies to ensure consistency. It is therefore proposed to compare the results of two examinations at 1.5 and 3 Tesla obtained on the same day on a series of 80 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years of age or older;
* Having an MRI indication of iron and fat quantification;
* Benefiting from social security;
* Having given a free, informed and written consent.

Exclusion Criteria:

Related to MRI

* Implantable cardiac pacemaker or defibrillator;
* Non-MRI cardiac valve compatible;
* Clips, stents, coils, etc ... no MRI compatible;
* Cochlear implants;
* Neuronal or peripheral stimulator;
* Foreign bodies metallic intra orbital or encephalic, foreign body close to the eyes, wound by metallic lash (war, ball);
* Endoprostheses placed for less than 4 weeks and osteosynthesis materials placed less than 6 weeks old;
* Claustrophobia;
* Pumps, tattoos, permanent make-up, intrauterine device, patches;
* Metallic, magnetic, non-removable material and close to the analysis field.

Other criteria

* unstable hemodynamic status, acute respiratory failure, general precarious condition or a need for continuous monitoring incompatible with MRI constraints;
* Persons subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty.
* Known pregnancy, breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Study of the agreement of the measurement of the fat and iron obtained by MRI, based on our previous calibrations (MRQuantif software), on two MRI devices. | Day 1
  Bland and Altman method comparing the quantification of iron and liver fat provided by the two MRI devices in the same patient using the MRQuantif software developed by the imaging department of the University Hospital of Rennes :
  * a 1.5 Tesla device
  * a 3 Tesla device

SECONDARY OUTCOMES:
Study of the concordance of the estimation of the quantification of the iron and the hepatic fat provided by our method and those of the constructors | Day 1
  Concordance of the estimation of the quantification of the iron and the hepatic fat provided by our method and those of the constructors
Analysis of the repeatability of the measurement (two acquisitions for each study). | Day 1
  Intraclass correlation coefficients (ICCs) and Bland & Altmann between two acquisitions
Analysis of the intra or interobserver reproducibility (several analysis for a single acquisition). | Day 1
  Intraclass correlation coefficients (ICCs) and Bland & Altmann between two readers/readings

CONTACTS AND LOCATIONS:
Overall Officials: Yves Gandon, MD, PhD, Principal Investigator — Rennes University Hospital
Locations (2):
- France (2):
  - Hôpital St Vincent du Groupement des Hôpitaux de l'Institut Catholique de Lille, Lille
  - CHU de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No